CLINICAL TRIAL: NCT04193956
Title: Towards Patient-tailored Cancer Immunotherapy Supported by a Multifaceted Predictive Signature Composed of Integrative Omics and Molecular Imaging
Brief Title: POINTING: Clinical Cohort Study of Patients With Melanoma and NSCLC Receiving Checkpoint Inhibitors
Acronym: POINTING
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: POINTING
Record Dates: First submitted 2018-09-24; First posted 2019-12-11 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Melanoma; Non-Small Cell Lung Cancer
Keywords: Immunotherapy; Anti-PD1 checkpoint inhibitor
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsies, venous blood samples, feces samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- POINTING
  Interventions: Other: Standard-of-care procedures; Other: Study procedures

INTERVENTIONS:
Other: Standard-of-care procedures — Patients receive standard of care anti-PD-1 treatment as monotherapy or in combination with other checkpoint inhibitors. Related assessments, as laboratory assessments, CT-thorax-abdomen and FDG-PET will be performed according to clinical routine procedures.
Other: Study procedures — Patients will undergo tumor biopsies, venous blood sampling and feces sampling in combination with a food questionnaire before, during and at the end of standard of care anti-PD-1 treatment.

SUMMARY:
This is a two-center, prospective continuously accruing longitudinal cohort study in patients with non-small cell lung carcinoma (NSCLC) or metastatic melanoma eligible for standard anti-PD-1 antibody treatment. The data from this prospective longitudinal cohort will be used in the POINTING (towards patient -tailored cancer immunotherapy supported by a multifaceted predictive signature composed of integrative omics and molecular imaging) KWF Kankerbestrijding project (WP4). The goal of this project is to develop a multifaceted predictive signature, by using new techniques on tumor characteristics before and during treatment with immune therapy. To do so, researchers will use the 'omics' approach. By combining molecular omics comprising genomics, transcriptomics, proteomics with radiomics and molecular imaging a set of factors will arise which can accurately predict the outcome of the treatment.

Participants in this cohort will undergo tumor biopsies, venous blood sampling and feces sampling before, during and at the end of standard anti-PD-1 antibody treatment. Also, data derived form routine procedures performed for standard-of-care anti-PD-1 treatment (ao laboratory assessments, CT and FDG-PET) will be collected.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytological documented locally advanced or metastatic melanoma or NSCLC.
2. Patients must be eligible for standard treatment with anti-PD-1 antibody treatment (monotherapy or in combination with other checkpoint inhibitors).
3. Age ≥18 years.
4. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions.
5. Metastatic or locally advanced lesion(s) of which a histological biopsy can safely be obtained according to standard clinical care procedures.
6. Ability to comply with protocol.
7. Signed Informed Consent form.

Exclusion Criteria:

1. Malignancies other than melanoma or NSCLC within 5 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent or ductal carcinoma in situ treated surgically with curative intent).
2. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to study inclusion.

   * Patients who have received acute, low-dose, systemic immunosuppressant medications may be enrolled.
   * The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g. fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic melanoma or metastatic NSCLC, who are eligible to receive anti-PD-1 antibody treatment as monotherapy or in combination with other checkpoint inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Predictive signatures based on multi-omics for PD-1 antibody treatment response as assessed by RECIST1.1 | 5 years
  The aim of this clinical cohort is to develop and validate multifaceted predictive signatures for PD-1 antibody effects with relevant components of integrative omics (histology, immunohistochemistry, genomics, transcriptomics, proteomics, radiomics and/or molecular imaging), which predict, which patients have a ≤ 5% chance of responding to anti-PD-1 antibody treatment.

SECONDARY OUTCOMES:
2. Predictive signatures based on multi-omics for PD-1 antibody treatment toxicity as assessed by CTCAE 4.03. | 5 years
  As secondary aim, the relation between multifaceted signatures composed by relevant components of integrative omics (histology, immunohistochemistry, genomics, transcriptomics, proteomics, radiomics and/or molecular imaging) and toxicity of PD-1 antibody treatment will be assessed. Toxicity will be scored according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: E. G.E. de Vries, MD, PhD, Study Chair — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - NKI-AvL, Amsterdam
  - University Medical Center Groningen, Groningen